CLINICAL TRIAL: NCT02642406
Title: Safety, Efficacy and Patient Reported Outcomes of Advanced Breast Cancer Patients: Therapy Management With Nab-Paclitaxel in Daily Routine - SERAPHINA
Brief Title: Therapy Management With Nab-Paclitaxel in Daily Routine
Acronym: SERAPHINA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: SEN2015-01
Record Dates: First submitted 2015-12-09; First posted 2015-12-30 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Despite treatment improvements in breast cancer, a large number of patients still progress to the metastatic stage. Metastatic breast cancer patients have an extremely unfavorable prognosis. Not only efficacy, but also quality of life are in the focus when planning a therapy or therapy sequence for metastatic breast cancer patients. Therapy options include anti-hormonal Therapy, antibody therapies, other targeted therapies and chemotherapies. One of the most effective chemotherapies in the adjuadjuvant and metastatic setting is paclitaxel. However drug handling and its side effects can compromise patients quality of life and can have an impact on the pharmacokinetics of the drug.

In metastatic breast cancer patients increasing therapy efficacy and reduction of side effect frequency are considered to be advancements of therapy. One of these advancements is the development of a cremophor free and albumin bound paclitaxel, nab-Paclitaxel (Abraxane), which is thought to have a better efficacy and reduced toxicity profile. Nab-Paclitaxel is approved for the treatment of metastatic breast cancer after a failure of first-line therapy and when antracyclines are not indicated.

The SERAPHINA study aims to investigate in the use of nab-Paclitaxel in daily routine and the frequency and perception of side effects.

As a non-interventional study, the SERAPHINA Study will assess the patient characteristics and describe the patient cohort, in which nab-Paclitaxel is given. This includes age distribution and characteristics documented by the patients themselves.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer in which a therapy with nab-paclitaxel was indicated by the treating physician
* Treatment of nab-Paclitaxel must either have not been started yet, or first application of nab-Paclitaxel was not prior to 21 days before study entry
* Female patients, age ≥18 years
* Invasive breast cancer (irrespective of status of BC, e.g. TNM, receptor status etc.)
* Metastatic or locally advanced, inoperable disease proven by clinical measures (i.e. standard imaging)
* Patients scheduled for nab-Paclitaxel treatment in daily routine before screening
* Patients, who are able and willing to sign the informed consent form

Exclusion Criteria:

* Patient is currently enrolled, or will enroll in an interventional clinical study in which investigational therapeutic procedures are performed or investigational therapies are administered while participating in this study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1200 patients with locally advanced/metastatic breast cancer for who is curruently or will be treated with nab-Paclitaxel according to the approval as stated in the Summary of Product Characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2015-12; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Epidemiological assessment of progression free survival (PFS) under real life conditions. | A patient remains in the study for a maximum of 36 months or until death, whatever occurs first
  PFS defined as the time to the first progression or death after therapy start of nab-Paclitaxel.

SECONDARY OUTCOMES:
Assessment of other prognostic characteristics | A patient remains in the study for a maximum of 36 months or until death, whatever occurs first
  OS (overall survival) is defined as the time to death from therapy start of nab-Paclitaxel. Reason for death is taken into consideration as well (BBCS, breast cancer specific survival).
Influence of age on the prognosis and quality of life. | A patient remains in the study for a maximum of 36 months or until death, whatever occurs first
  Progression free survival, overall survival and quality of life assessed with PRO
Incidence of adverse events, serious adverse events will be reported. | A patient remains in the study for a maximum of 36 months or until death, whatever occurs first
  NCI Common Toxicity Criteria Version 4.03
Quality of life (FACT-B -Taxane, Version 4, nab-Paclitaxel specific questions, NCCN-Distress-Thermometer) | A patient remains in the study for a maximum of 36 months or until death, whatever occurs first
  Patient reported (PRO) quality of life is assessed with standardized questionnaires (FACT-B, Version 4, FACT-Taxane, Version 4, nab-Paclitaxel specific questions, NCCN-Distress-Thermometer.
Influence of breast cancerpatient characteristics on prognosis, adverse event frequencies, quality of life and therapy decision making. | A patient remains in the study for a maximum of 36 months or until death, whatever occurs first
  The patient group is described by patient and tumor characteristics and a series of questionnaires assessing health and socioeconomic status and geriatric assessment status. These parameters that describe the patient cohort will be analyzed with regard to their influence on prognosis, adverse event frequencies, quality of life and therapy decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fasching, Prof. Dr., Principal Investigator — Frauenklinik des Universitätsfrauenklinikums Erlangen; Hans Joachim Lück, Prof. Dr., Principal Investigator — Gynäkologisch-Onkologische Schwerpunktpraxis am Pelikanplatz; Diethelm Wallwiener, Prof. Dr., Study Director — Universitätsklinikum Tübingen Universitäts-Frauenklinik; Sara Brucker, Prof. Dr., Study Director — Universitätsklinikum Tübingen Universitäts-Frauenklinik
Locations (83):
- Germany (83):
  - Aalen Brustzentrum, Aalen, Baden-Wurttemberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - NCT Heidelberg, Heidelberg, Baden-Wurttemberg
  - Frauenklinik des Städtischen Klinikums, Karlsruhe, Baden-Wurttemberg
  - St. Vicentius Kliniken gAG, Karlsruhe, Baden-Wurttemberg
  - Ortenau Klinikum Lahr-Ettenheim, Lahr, Baden-Wurttemberg
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Paracelsus Krankenhaus Ruit, Ruit, Baden-Wurttemberg
  - Schwerpunktpraxis für Hämatologie und Internistische Onkologie, Gastroenterologie, Singen, Baden-Wurttemberg
  - Brustzentrum, Stuttgart, Baden-Wurttemberg
  - Universitätsfrauenklinik Tübingen, Tübingen, Baden-Wurttemberg
  - GRN-Klinik Weinheim Abteilung für Gynäkologie und Geburtshilfe, Weinheim, Baden-Wurttemberg
  - Klinikum für Frauenheilkunde und Geburtshilfe Esslingen, Esslingen am Neckar, Baden-Württenberg
  - MVZ Amberg, Amberg, Bavaria
  - phase drei Hämato-Onkologischer Studienkreis am Klinikum Aschaffenburg, Aschaffenburg, Bavaria
  - Klinikum Augsburg Frauenklinik, Augsburg, Bavaria
  - Sozialstiftung Bamberg, Klinikum am Bruderwald Klinik für Frauenheilkunde und Geburtshilfe, Bamberg, Bavaria
  - Sozialstiftung Bamberg, Klinikum am Bruderwald Klinik für Frauenheilkunde und Geburtshilfe, Bayreuth, Bavaria
  - Rottal-Inn-Kliniken GmbH, Eggenfelden, Bavaria
  - Universitätsfrauenklinik Erlangen, Erlangen, Bavaria
  - Praxis für Hämatologie Onkologie Palliativmedizin, Landshut, Bavaria
  - Praxisgemeinschaft Dr. med. Steffi Busch, Mühlhausen, Bavaria
  - MOPS Elisenhof MOP-Studiengesellschaft, München, Bavaria
  - Klinikum der Universität München (LMU), München, Bavaria
  - Praxisgemeinschaft - Frauenärzte am Stadtpark, Nuremberg, Bavaria
  - Caritas-Krankenhaus St. Josef, Regensburg, Bavaria
  - MVZ Weiden GmbH, Weiden, Bavaria
  - Praxis Dr. med. Uwe G. Pöhls und Kollegen Fachärzte für Frauenheilkunde und Geburtshilfe, Würzburg, Bavaria
  - Onkologische Gemeinschaftspraxis, Würzburg, Bavaria
  - Akad. Lehrkrankenhaus der Charité, Ludwigsfelde, Brandenburg
  - Ruppiner Kliniken GmbH, Neuruppin, Brandenburg
  - g.SUND Gynäkologie Kompetenzzentrum, Stralsund, Brandenburg
  - Brustzentrum am Elisabeth-KH Leipzig, Leipzig, Dresden
  - Klinikum Darmstadt, Darmstadt, Hesse
  - Zentrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main, Hesse
  - Agaplesion Markus Krankenhaus, Frankfurt am Main, Hesse
  - MVZ Onkologische Kooperation Harz, Goslar, Hesse
  - Praxis Ammon/Meyer, Göttingen, Hesse
  - Klinikum Kassel GmbH, Kassel, Hesse
  - Frauenklinik Wetzlar, Wetzlar, Hesse
  - Niels-Stensen-Kliniken, Georgsmarienhütte, Lower Saxony
  - Gynäkologisch-Onkologische Praxis am Pelikanplatz, Hanover, Lower Saxony
  - Klinik f. Frauenheilkunde u. Geburtshilfe, Hanover, Lower Saxony
  - Frauenarzt Bewer und Sternberg Gynäkologie, Hanover, Lower Saxony
  - Gemeinschaftspraxis f. Hämatologie u. Onkologie, Westerstede, Lower Saxony
  - Facharztzentrum am Schloß, Wolfenbüttel, Lower Saxony
  - Evangelisches Krankenhaus Bethedsa Mönchengladbach GmbH, Mönchengladbach, Nordrhein-Westfalens
  - MarienHospital Onkologische Praxis, Bonn, North Rhine-Westphalia
  - Marienhospital Bottrop gGmbH, Bottrop, North Rhine-Westphalia
  - Gemeinschaftspraxis f. Onkologie und Hämatologie, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln g.GmbH, Cologne, North Rhine-Westphalia
  - Universitätsfrauenklinik Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - PIOH Praxis Internistischer Onkologie und Hämatologie, Frechen, North Rhine-Westphalia
  - Dokusan Gesellschaft für medizinische studien mbH & Co .KG, Herne, North Rhine-Westphalia
  - Helios Klinikum Krefeld, Krefeld, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Marienkrankenhaus/Brustzentrum, Schwerte, North Rhine-Westphalia
  - Praxisnetzwerk Hämatologie/Onkologie, Troisdorf, North Rhine-Westphalia
  - Onkologische Praxis, Velbert, North Rhine-Westphalia
  - Fachinternistische Gemeinschaftspraxis, Witten, North Rhine-Westphalia
  - Hämatologisch-Onkologische Praxis Würselen, Würselen, North Rhine-Westphalia
  - Schwerpunktpraxis für Hämatologie und Onkologie Hansen/Reeb/Pfitzner-Dempfle/Stehle, Kaiserslautern, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Poliklinik Chemnitz GmbH, Chemnitz, Saxony
  - Onkozentrum Dresden, Dresden, Saxony
  - Onkologische Gemeinschaftspraxis Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Klinikum Obergöltzsch Rodewisch, Rodewisch, Saxony
  - KKH Torgau, Brustzentrum, Torgau, Saxony
  - Johanniter-Krankenhaus Genthin-Stendal Klinik für Frauenheilkunde und Geburtshilfe, Stendal, Saxony-Anhalt
  - Christian-Albrecht-Universitäts Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Gynäkologische Gemeinschaftspraxis, Berlin
  - Charité, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Gynäkologische Praxisklinik Harburg, Hamburg
  - Praxis für Frauen, Ilsede
  - Universitätsklinikum Münster, Münster
  - Haveland Kliniken GmbH, Nauen
  - MVZ Kloster Paradiese GbR, Soest
  - Schwerpunktpraxis Onkologie, Speyer

IPD SHARING:
Plan to Share IPD: Undecided